CLINICAL TRIAL: NCT04338308
Title: New-generation Drug Eluting Stent vs. Bare Metal Stent in Saphenous Vein Graft - 1 Year Outcomes by a Propensity Score Ascertainment (SVG Baltic Registry)
Brief Title: New-DES vs BMS in SVG -1 Year Outcomes
Acronym: BALTIC
Status: Completed | Type: Observational
Sponsor: Medical University of Silesia (Other)
Collaborators: Wojciech Wojakowski (Unknown)
Responsible Party: Principal Investigator, Wojciech Wańha, MD, PhD, Medical University of Silesia
Other Study IDs: 01
Record Dates: First submitted 2020-04-04; First posted 2020-04-08 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Coronary Artery Disease
Keywords: Percutaneous coronary intervention; Saphenous vein graft; New generation drug-eluting stent; Bare metal stent
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SVG PCI
  Interventions: Device: new-DES; Device: BMS

INTERVENTIONS:
Device: new-DES — with ot without embolic protection device
Device: BMS — with ot without embolic protection device

SUMMARY:
Data regarding the efficacy of the percutaneous coronary intervention (PCI) with new-designed drug-eluting stent (new-DES) vs. bare metal stent (BMS) of saphenous vein grafts (SVG) stenosis is scarce. The primary objective was to compare one-year clinical outcomes of PCI in stenosis of SVG using new-DES vs. BMS in a real-world population. We carried out a multi-center registry comparing new-DES with BMS in all consecutive patients undergoing PCI of SVG. The primary composite endpoint was major adverse cardiac and cerebrovascular events (MACCE) at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* patients after CABG with significant SVG stenosis referred for PCI

Exclusion Criteria:

* patients who had both types of stents implanted in the same procedure
* patients with the old-DES
* patients who had PCI of other vascular territories during the same procedure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients undergoing PCI of SVG
Sampling Method: Non-Probability Sample
Enrollment: 792 (Actual)
Dates: Start 2008-02-01 (Actual); Primary Completion 2015-10-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
major adverse cardiac and cerebrovascular event | 1 year

SECONDARY OUTCOMES:
death | 1 year
myocardial infarction | 1 year
target vessel revascularization | 1 year
target lesion revascularization | 1 year
stroke | 1 year

CONTACTS AND LOCATIONS:
Locations (3):
- Poland (3):
  - First Department of Cardiology, Medical University of Gdansk, Gdansk, Poland, Gdansk
  - Department of Cardiology and Structural Heart Diseases, Medical University of Silesia, Katowice, Poland, Katowice
  - Second Department of Cardiology, Jagiellonian University Medical College, Krakow, Poland, Krakow

REFERENCES:
- [Background] Wanha W, Mielczarek M, Roleder T, Ladzinski S, Milewski M, Gilis-Malinowska N, Chmielecki M, Ciecwierz D, Bachorski W, Kunik P, Trznadel A, Mecka K, Genc A, Januszek R, Paczek P, Dziewierz A, Bartus S, Gruchala M, Smolka G, Dudek D, Navarese EP, Ochala A, Jaguszewski M, Wojakowski W. New-generation drug eluting stent vs. bare metal stent in saphenous vein graft - 1 year outcomes by a propensity score ascertainment (SVG Baltic Registry). Int J Cardiol. 2019 Oct 1;292:56-61. doi: 10.1016/j.ijcard.2019.04.022. Epub 2019 Apr 11. PMID 31003797